CLINICAL TRIAL: NCT02775773
Title: Longitudinal Clinical, Controlled, Randomized, Open-label, Phase III Study to Assess the Equivalence of Tranexamic Acid (TXA) vs Oxytocin (OXY) in Reducing Post Partum Haemorrhage (PPH) in Patients at the End of Pregnancy (37-42 w), at Low Risk of PPH
Brief Title: Clinical Study to Assess the Equivalence of Tranexamic Acid vs Oxytocin in Reducing the PPH
Acronym: TRANOXY2016
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda U.S.L. 1 di Massa e Carrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Azenda USLToscana Nord Ovest
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2019-01

CONDITIONS: Post Partum Haemorrhage
Keywords: TXA; PPH
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm A (TXA) (Experimental): 2 vials (=1 gram ) of Tranexamic Acid administered slow intravenous infusion within 5 minutes from the delivery(third stage after labor)
  Interventions: Drug: Tranexamic Acid
- arm B (OXY) (Active Comparator): 2 vials (=10 IU/International Unit) of oxytocin administered intramuscularly within 5 minutes from the delivery (third stage after labor)
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Tranexamic Acid — 2 vials ( =1 gram) of Tranexamic Acid slow intravenous infusion administered within 5 minutes from the delivery (third stage after labor)
  Other Names: TXA
  Arms: arm A (TXA)
Drug: Oxytocin — 2 vials (=10 IU/International Unit) of Oxytocin administered intramuscularly within 5 minutes from the delivery (third stage after labor)
  Other Names: OXY
  Arms: arm B (OXY)

SUMMARY:
The purpose of this study was to evaluate that the tranexamic acid (TXA)Intravenous and oral, is equivalent oxytocin (OXY),intramuscularly, in reducing the blood loss in post partum period (mL) in patients at the end of pregnancy ( 37-42 w ) at low risk of post partum hemorrhage (PPH). The PPH means a blood loss equal to or greater than 500 ml after a vaginal delivery (the bleeding is defined severe if it exceeds 1000 mL). PPH is called "primary" when blood loss arose within 24 hours after birth.

DETAILED DESCRIPTION:
This trial includes three arms of treatment :

* arm A (IMP1Test): TXA 500 mg/ 2 vials (1 gr) slow intravenous infusion 1ml/min within 5 minutes from the delivery(third stage af labor)
* arm B (IMP2Control): OXY 5 IU/ml/ 2 vials (10 International Unit) intramuscularly within 5 minutes from the delivery (third stage af labor) The clamping of the umbilical cord will be executed immediately after birth.

The randomization 1:1 (block design), generated by the computer.

Primary outcomes: assessment of total blood loss expressed in mL:

* immediately after delivery
* two hours after delivery

The measurement of the overall blood loss at delivery (ml) will be performed by the graduated bag, immediately after birth.

The measurement two hours after delivery will be performed by weighing of the adsorbent material [ N.ml = N. gr indicated by the balance - dry weight of the sanitary napkin]. The overall loss in blood measured (ml) two hours of delivery will then be performed by adding the two collections.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at the end of pregnancy ( 37-42 w ) at low risk of PPH Mean by low-risk of PPH subjects without any of the following risk factors : hypertension/preeclampsia, placental abruption during pregnancy , placenta previa , tocolysis two hours before delivery, multiple pregnancy , previous PPH, obesity ( BMI > 35 ), anemia (Hb < 7 g/dL), elective caesarean section , induction of labor, retention of placental material , polyhydramnios , fever during labor, use of high doses of heparin low molecular weight.
* Subjects full capacity and the willingness to give written informed consent .

Exclusion Criteria:

* Subjects with preterm pregnancy (<37 weeks ) or with prolonged pregnancy ( > 42 weeks )
* Subjects at the end of pregnancy ( 37 weeks - 42 weeks ) with the following risk factors for PPH (Tab1.Protocol Study, vers.2.0 of 07/05/2016)
* multiple pregnancy
* History of thromboembolic disease or high incidence of thromboembolic events in family history ( patients at high risk of thrombophilia )
* Patients with Long - QT syndrome or who are taking drugs that cause QT prolongation
* Intrauterine fetal Death
* Epilepsy
* Autoimmune disease Tab1 medical history :
* Placental abruption during pregnancy
* Placenta previa
* Hypertension / preeclampsia
* Previous PPH
* Polyhydramnios
* Obesity ( BMI > 35 )
* Anemia ( < 7 g / dL )

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 256 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
assessment of total blood loss expressed in mL | immediately after delivery
  global blood loss > 500 mL
assessment of total blood loss expressed in mL | two hours after delivery
  global blood loss > 500 mL

SECONDARY OUTCOMES:
assessment of the number of hemodynamic changes | two hours after delivery
  hypotension (number of women with Arterial Pressure < 100/60 mm/Hg )
assessment of the number of hemodynamic changes | immediately after delivery
  increased heart rate (number of women with Heart Rate > 60 bpm )
assessment of the need of using additional uterotonic | immediately after delivery
  administration additional drug for the treatment of PPH
assessment of the need of using additional uterotonic | two hours after delivery
  administration additional drug for the treatment of PPH
assessment the need for surgical manoeuvres for the bleeding control | immediately after
  need of intrauterine balloon or uterine compression sutures for surgical treatment of the PPH or hysterectomy
assessment the need for surgical manoeuvres for the bleeding control | two hours after
  need of intrauterine balloon or uterine compression sutures for surgical treatment of the PPH or need of intrauterine balloon or uterine compression sutures for surgical treatment of the PPH or hysterectomy
assessment the need for the blood transfusions | two days after delivery
  Hb <7 g/dL
evaluation of the number of cases in which the following was seen verified: | two days after delivery
  nausea between delivery and discharge vomiting between birth and discharge headache between birth and discharge dyspnoea between birth and discharge Chest pain between birth and discharge endometritis after delivery (assessed by monitoring body temperature)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ostetricia e Ginecologia-Ospedale delle Apuane, Massa, MS, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ragusa A, Ficarola F, Ferrari A, Spirito N, Ardovino M, Giraldi D, Stuzziero E, Rinaldo D, Procaccianti R, Larciprete G, De Luca C, D'Avino S, Principi G, Angioli R, Svelato A. Tranexamic acid versus oxytocin prophylaxis in reducing post-partum blood loss, in low-risk pregnant women: TRANOXY STUDY, a phase III randomized clinical trial. EClinicalMedicine. 2024 May 31;73:102665. doi: 10.1016/j.eclinm.2024.102665. eCollection 2024 Jul. PMID 38873634